CLINICAL TRIAL: NCT06097923
Title: Implementation of Fluid Strategies Using Real-time Bioelectrical Analyzer of Postoperative Patients in Surgical Intensive Care Unit (SICU); a Novel Guidance to Set an Ideal Fluid Status of Patient in Acute Postoperative Phase
Brief Title: Implementation of Fluid Strategies Using Real-time Bioelectrical Analyzer in Surgical Intensive Care Unit (SICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Eun Young Kim, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIA_03
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Fluid Overload; Fluid Loss
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active fluid management with BIA monitoring (Experimental): For assessment of fluid status, a commercial portable BIA device (InBody M20®, InBody Corp., Seoul, Korea) was measured. Baseline BIA data were collected at the time of ICU admission, and BIA measurements were performed daily for 3days for all participants. The participants in active fluid management with BIA monitoring arm received fluid supplementation targeting specific range of ECW ratio by BIA (0.390-0.406). If a patient with dehydrated status indicated by the ECW ratio was less than 0.390, a bolus infusion was performed using 250ml of crystalloid fluid (PlasmaLyte). If a patient with overhydrated status indicated by the ECW ratio was more than 0.406, 10mg of furosemide was administered. Changes in the ECW ratio were measured at one hour after initial intervention for fluid adjustment, and the investigators determined whether additional intervention was needed according to results of changes. These processes continued until the ECW ratio was within the normal range (0.390-0.406).
  Interventions: Drug: Active fluid management with BIA monitoring
- Conventional fluid management without BIA monitoring (Experimental): For assessment of fluid status, a commercial portable BIA device with 5-kilohertz, 50-kilohertz, and 250-kilohertz alternating current (InBody M20®, InBody Corp., Seoul, Korea) was measured. Baseline BIA data were collected at the time of ICU admission. Thereafter, BIA measurements were performed daily for 3 days for all participants.
  The participants in conventional fluid management without BIA monitoring arm underwent conventional fluid management without specific targets of ECW ratio by BIA.
  Interventions: Drug: Conventional fluid management without BIA monitoring

INTERVENTIONS:
Drug: Active fluid management with BIA monitoring — The participants in active fluid management with BIA monitoring arm received fluid supplementation targeting specific range of ECW ratio by BIA (0.390-0.406). If a patient with dehydrated status indicated by the ECW ratio was less than 0.390, a bolus infusion was performed using 250ml of crystalloid fluid (PlasmaLyte). If a patient with overhydrated status indicated by the ECW ratio was more than 0.406, 10mg of furosemide was administered. Changes in the ECW ratio were measured at one hour after initial intervention for fluid adjustment, and these processes continued until the ECW ratio was within the normal range (0.390-0.406).
  Arms: Active fluid management with BIA monitoring
Drug: Conventional fluid management without BIA monitoring — The participants in conventional fluid management without BIA monitoring arm underwent conventional fluid management without specific targets of ECW ratio by BIA.
  Arms: Conventional fluid management without BIA monitoring

SUMMARY:
Precise assessment of postoperative volume status is important to administrate optimal fluid management. Bioelectrical impedance analysis (BIA) which measures the body composition using electric character. Extracellular water (ECW) ratio by BIA represented as the ratio of ECW to total body water (TBW) and is known to reflect the hydration status. Based on this, we aimed to determine whether aggressive fluid control using ECW ratio could improve clinical outcomes through a single blind, randomized controlled trial.

DETAILED DESCRIPTION:
Critically ill patients admitted to an intensive care unit (ICU) after surgery have commonly experienced a large amount of wide organ injury and profuse bleeding resulting in vessel damage during surgery. Severe systemic inflammatory reactions and pathophysiological stress could consequently occur in these patients. For patients in an acute postoperative phase, it is important to maintain organ perfusion by correcting hemodynamic instability through fluid resuscitation.

Bioelectrical impedance analysis (BIA), a non-invasive method, is useful for quantitatively measuring body composition such as body fat and muscle mass. It is also useful for evaluating volume status based on resistance and reactance of cells known to have different electrical conductivity according to biological characteristics of body composition. In our previous study using BIA, the results showed that changes in ECW ratio after surgery were related to conventional parameters of overhydrated status such as daily fluid balance or capillary leak index (CLI). In addition, overhydration with value of ECW ratio above 0.390 on 3rd postoperative day appeared to be a risk factor for postoperative morbidity and mortality.

Herein, we aim to set the ECW ratio as a guideline for postoperative volume status and confirm a hypothesis that active intervention with fluid management to control the ECW ratio by BIA could lower clinical outcomes in patients with fluid imbalance through a prospective randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the surgical ICU after surgery under general anesthesia regardless of the type of surgery
* Patients who showed abnormal range of baseline ECW ratio by BIA (less than 0.390 or more than 0.405) that measured at the time of ICU admission

Exclusion Criteria:

* aged under 18 years
* underwent surgery under local or regional anesthesia
* pregnant
* had bone fixation or underwent limb amputation
* had any prosthetic medical devices such as pacemaker or metallic intravascular device
* stayed in ICU for less than 48 hours
* readmitted within 48 hours after ICU discharge
* diagnosed with renal failure and receiving renal replacement therapy
* underwent extracorporeal membrane oxygenation treatment before surgery
* agreed for do-not-resuscitate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality rate | Participants were followed upto 28th day after surgery
  Proportion of patients who died during the hospitalization period among participants

SECONDARY OUTCOMES:
Incidence of postoperative morbidities | Participants were followed upto 28th day after surgery
  Proportion of patients who experienced postoperative complications among participants
28-day mortality rate | Participants were followed upto 28th day after surgery
  Proportion of patients who died within 28 days after surgery among participants

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Trauma and Surgical Critical Care, Department of Surgery, Seoul St. Mary's Hospital, Seoul, Seocho-gu, Banpo-dong Banpodaero 222, South Korea

REFERENCES:
- [Derived] Chung YJ, Lee GR, Kim HS, Kim EY. Effect of rigorous fluid management using monitoring of ECW ratio by bioelectrical impedance analysis in critically ill postoperative patients: A prospective, single-blind, randomized controlled study. Clin Nutr. 2024 Sep;43(9):2164-2176. doi: 10.1016/j.clnu.2024.07.040. Epub 2024 Jul 31. PMID 39142110